CLINICAL TRIAL: NCT06876415
Title: Monitoring of Occlusion Pressure and Esophageal Pressure to Guide Weaning From Venovenous ECMO in ARDS: a Randomized Controlled Study
Brief Title: Free for Weaning ECMO vs Respiratory Driven Study
Acronym: FORWARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RCAPHM23_0464; ID-RCB (Other: 2024-A01472-45)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: veno-venous ECMO; Decannulation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Investigator
Masking Description: P0.1 and delta Poeso values will be monitored in a blinded manner by an independent investigator and will not be integrated into the decannulation decision
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECMO-physio group (Experimental): Patients undergo the ultimate vvECMO weaning test with minimal ECMO support (ECMO flow ≤ 3 L/min, fresh gas flow ≤ 1 L/min, FiO2 21%) and mechanical ventilation with partial support, allowing spontaneous ventilation. P0.1 and delta Poeso values will be monitored and integrated into the decannulation decision
  Interventions: Other: P0.1 and delta Poeso integration into the decanulation decision
- ECMO-gazo group (No Intervention): Patients undergo the ultimate vvECMO weaning test with minimal ECMO support, similar to the experimental group. P0.1 and delta Poeso values will be monitored in a blinded manner by an independent investigator and will not be integrated into the decannulation decision.

INTERVENTIONS:
Other: P0.1 and delta Poeso integration into the decanulation decision — P0.1 and delta Poeso integration into the decanulation decision
  Arms: ECMO-physio group

SUMMARY:
In its most severe form, Acute Respiratory Distress Syndrome (ARDS) may require the use of veno-venous ECMO (vvECMO). While the criteria for vvECMO indication, ECMO settings, and ventilator management are relatively well-defined after the publication of the EOLIA trial and subsequent national or international guidelines, few studies have assessed the criteria and methods for weaning from vvECMO. Besides, advances in the understanding of the pathophysiology of mechanical ventilation (MV) weaning process have led to the development of specific monitoring tools for this phase.

Schematically, respiratory drive can be evaluated via the ventilator by measuring the pressure generated during a 100-millisecond expiratory occlusion (P0.1) and respiratory efforts through the measurement of esophageal pressure variation (delta Poeso).

Recent retrospective studies conducted on COVID-19 ARDS patients supported by vvECMO suggest a longer duration of mechanical ventilation for patients whose weaning and decannulation process was "forced," i.e., performed under conditions of significant respiratory drive and effort. High values of P0.1 and delta Poeso were associated with prolonged MV duration. Self-inflicted lung injury (P-SILI) and elevated transpulmonary pressure related to these uncontrolled respiratory efforts likely explain the negative impact on MV duration.

Therefore, this randomized study proposes to assess these monitoring tools, which are regularly used in clinical practice, to guide vvECMO weaning and decannulation decisions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older Patient whose trusted person has given consent for participation in the study
* Patient on veno-venous ECMO with weaning criteria, including:
* Resolution of the cause of ARDS
* Absence of hemodynamic instability, defined as norepinephrine dose ≤ 0.5 μg/kg/min for at least 3 hours
* Use of a ventilatory mode that allows spontaneous ventilation (VS-AI, BiPAP, or APRV)
* Maximum inspiratory pressure ≤ 28 cm H2O, with a maximum driving pressure ≤ 15 cm H2O, enabling tidal volumes between 4 and 8 ml/kg of predicted body weight (PBW)
* ECMO membrane sweep flow ≤ 2 L/min
* Patient protected by social security

Exclusion Criteria:

* Contraindication to the placement of an esophageal pressure balloon (e.g., esophageal varices, nasal trauma, uncontrolled coagulopathy, severe thrombocytopenia),
* Patient with treatment limitation at the time of inclusion,
* Patient in the time frame of exclusion from another research protocol at the time of consent signing,
* Vulnerable patients: minor, adult patient under guardianship or curatorship, patient deprived of liberty, pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation from ECMO decannulation to weaning from mechanical ventilation | 60 days after inclusion
  The weaning from mechanical ventilation is defined as the absence of mechanical ventilation for 48 consecutive hours.
P0.1 and delta Poeso measurements | From inclusion to 48h after decanulation
  P0.1 and delta Poeso values will be monitored and tracked at inclusion and then every 8 hours until decannulation, and up to 48 hours after decannulation.
  In the experimental group, these values will be incorporated into the criteria guiding the decannulation decision.
  In the control group, these values will be monitored and recorded by an investigator who is not involved in the decannulation decision. These values will not be included in the criteria guiding the decannulation decision.

SECONDARY OUTCOMES:
Mortality rate in intensive care unit | 60 days after inclusion
Mortality rate in hospital | 60 days after inclusion
Intensive care unit stay duration from inclusion | 60 days after inclusion
Hospital stay duration from inclusion | 60 days after inclusion
Total number of days spent on ECMO from admission to intensive care unit discharge | 60 days after inclusion
Total duration of mechanical ventilation | 60 days after inclusion
Time between the start of mechanical ventilation and ECMO cannulation | 60 days after inclusion
Number of ventilator-free days | 60 days after inclusion
Number of patients decannulated and then re-initiated on vvECMO | 60 days after inclusion
Number of patients requiring controlled ventilation for at least 24 hours after decannulation | 60 days after inclusion
Number of days with continuous sedation with or without continuous paralysis after decannulation | 60 days after inclusion
Incidence of barotrauma assessed by radiographs and clinical examination after decannulation | 60 days after inclusion
Percentage of patients placed in prone positioning after decannulation | 60 days after inclusion
Number of days on inhaled nitric oxide after decannulation | 60 days after inclusion
Neuromyopathy on the day of decannulation | Day of decanulation
  Neuromyopathy will be assessed using the Medical Research Council score. Total score ranges from 0 (complete tetraplegia) to 60 (normal muscle strength).
Neuromyopathy on the day of weaning from mechanical ventilation | Day of weaning from mechanical ventilation
  Neuromyopathy will be assessed using the Medical Research Council score. Total score ranges from 0 (complete tetraplegia) to 60 (normal muscle strength).
Number of patients who received corticosteroid therapy | 60 days after inclusion
  ≥ 0.5 mg/kg of equivalent methylprednisolone

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (4):
- France (4):
  - Hospices Civiles de Lyon, Lyon
  - Assistance - Publique Hôpitaux de Marseille, Marseille
  - CHU de Nice, Nice
  - Assistance Publique - Hôpitaux de Paris, Paris

IPD SHARING:
Plan to Share IPD: No